CLINICAL TRIAL: NCT06638827
Title: Outcome of Bilateral Thoracoscopic Sympathectomy for Patients with Primary Focal Hyperhidrosis, Sohag University Hospital Experience
Brief Title: Outcome of Bilateral Thoracoscopic Sympathectomy for Patients with Primary Focal Hyperhidrosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mohamed Ashraf Mokhtar, Resident physician, Cardiothoracic Surgery department, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Soh-Med-24-09-09MS
Record Dates: First submitted 2024-10-06; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Hyperhidrosis Primary Focal Palms
Keywords: Hyperhidrosis; Primary focal hyperhidrosis
MeSH Terms: conditions — Hyperhidrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients complaining of primary focal hyperhidrosis (Active Comparator): This is a prospective clinical study that includes all patients with Primary Focal Hyperhidrosis, who will be operated on with Bilateral Thoracoscopic Sympathectomy.
  Interventions: Procedure: Thoracic Sympathectomy

INTERVENTIONS:
Procedure: Thoracic Sympathectomy — Bilateral thoracoscopic sympathectomy will be performed with general anesthesia, using single lung ventilation and monopolar cautery for transection of the sympathetic chain.
  Persons with PFH who underwent the BTS were classified into three groups, depending the level of transaction of sympathetic chain:
  1. transection at the level from the second to the forth thoracic sympathetic ganglion (T2- T4);
  2. transection at the level from the third to the forth thoracic sympathetic ganglion (T3-T4)
  3. transection at the level from the second to the third thoracic sympathetic ganglion (T2-T3)..
  Other Names: Bilateral Thoracoscopic Sympathectomy

SUMMARY:
The goal of this clinical trial is to examine the overall efficiency of Bilateral Thoracoscopic Sympathectomy on the permanent reduction of Primary focal hyperhidrosis of predilective parts of the body, palms, armpits, face, and soles.

DETAILED DESCRIPTION:
The aims of this study are:

1. examine the efficiency of Bilateral Thoracoscopic Sympathectomy (BTS) with different levels of transection among the persons with the Primary focal Hyperhidrosis (PFH)
2. examine the influence of BTS on cardio-pulmonary function tests in persons with PFH after the operation.
3. examine the incidence, duration, and intensity of compensatory sweating after BTS among persons with PFH
4. examine the incidence, duration, localization, and treatment of postoperative pain after BTS among persons with PFH.
5. determine postoperative complications of BTS among persons with PFH
6. examine the influence of BTS on quality of life among persons with PFH

ELIGIBILITY:
Inclusion Criteria:

* a. persons with confirmed and estimated Primary Focal Hyperhidrosis accepted to participate in this investigation, fulfilling pre and postoperative questionnaires about BTS effects and quality of life after the operation
* b. Satisfactory CardioPulmonary Function

Exclusion Criteria:

* previous thoracic surgical procedures, rib fractures, massive pneumonias, or pleural empyema
* Secondary Hyperhidrosis

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Reduction in Hyperhidrosis Severity as Assessed by the Hyperhidrosis Disease Severity Scale (HDSS) and Gravimetric Sweat Testing | Immediately After surgery
  Participants will be assessed using the HDSS and gravimetric sweat testing. A reduction of ≥ 2 points in HDSS score or a ≥ 50% reduction in sweat production will be considered a successful outcome. Data will be aggregated as the proportion of participants achieving these reductions.

SECONDARY OUTCOMES:
Change in Quality of Life as Assessed by the Dermatology Life Quality Index (DLQI) | From baseline to 3 months post-operation.
  The DLQI will be administered preoperatively and at 3 months postoperatively to evaluate changes in quality of life. The DLQI is a 10-item questionnaire where higher scores indicate greater impairment. The primary endpoint will be the mean reduction in DLQI score from baseline to 3 months, with a reduction of ≥ 5 points considered clinically significant
Postoperative Pain Levels as Measured by the Visual Analog Scale (VAS) | From 1 day post-operation to 1 month post-operation.
  Postoperative pain will be assessed at regular intervals (1 day, 1 week, and 1 month post-surgery) using the Visual Analog Scale (VAS), a 10-point scale where 0 indicates no pain and 10 indicates severe pain. The primary endpoint will be the mean VAS score at each time point, with pain reduction over time compared
Incidence and Severity of Compensatory Sweating as Measured by the Hyperhidrosis Disease Severity Scale (HDSS) | from time of operation for 3 months after operation
  Participants will report compensatory sweating at 1 month and 3 months post-surgery using the HDSS. The severity of compensatory sweating will be recorded with a scale ranging from 1 (no symptoms) to 4 (severe symptoms that interfere with daily activities). The primary endpoint will be the percentage of patients reporting compensatory sweating and their scores on the HDSS at 3 months
Incidence and Severity of Compensatory Sweating as Measured by the Hyperhidrosis Disease Severity Scale (HDSS) | From baseline to 3 months post-operation.
  Participants will report compensatory sweating at 1 month and 3 months post-surgery using the HDSS. The severity of compensatory sweating will be recorded with a scale ranging from 1 (no symptoms) to 4 (severe symptoms that interfere with daily activities). The primary endpoint will be the percentage of patients reporting compensatory sweating and their scores on the HDSS at 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University, Sohag, Sohag Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hornberger J, Grimes K, Naumann M, Glaser DA, Lowe NJ, Naver H, Ahn S, Stolman LP; Multi-Specialty Working Group on the Recognition, Diagnosis, and Treatment of Primary Focal Hyperhidrosis. Recognition, diagnosis, and treatment of primary focal hyperhidrosis. J Am Acad Dermatol. 2004 Aug;51(2):274-86. doi: 10.1016/j.jaad.2003.12.029. No abstract available. PMID 15280848
- [Background] Doolabh N, Horswell S, Williams M, Huber L, Prince S, Meyer DM, Mack MJ. Thoracoscopic sympathectomy for hyperhidrosis: indications and results. Ann Thorac Surg. 2004 Feb;77(2):410-4; discussion 414. doi: 10.1016/j.athoracsur.2003.06.003. PMID 14759407
- [Background] Shabat S, Furman D, Kupietzky A, Srour B, Mordechai-Heyn T, Grinbaum R, Mazeh H, Mizrahi I. Long-term Outcomes of Endoscopic Thoracoscopic Sympathectomy for Primary Focal Palmar Hyperhidrosis: High Patient Satisfaction Rates Despite Significant Compensatory Hyperhidrosis. Surg Laparosc Endosc Percutan Tech. 2022 Dec 1;32(6):730-735. doi: 10.1097/SLE.0000000000001100. PMID 36130719
- [Background] Milanez de Campos JR, Kauffman P, Gomes O Jr, Wolosker N. Video-Assisted Thoracic Sympathectomy for Hyperhidrosis. Thorac Surg Clin. 2016 Aug;26(3):347-58. doi: 10.1016/j.thorsurg.2016.04.010. PMID 27427529
- [Background] Solish N, Wang R, Murray CA. Evaluating the patient presenting with hyperhidrosis. Thorac Surg Clin. 2008 May;18(2):133-140. doi: 10.1016/j.thorsurg.2008.01.002. PMID 18557587